CLINICAL TRIAL: NCT06020638
Title: Determining The Effects Of Nasopharyngeal Suction With Negative And Positive Pressure: Randomised Conrolled Trial
Brief Title: Determining The Effects Of Nasopharyngeal Suction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Rukiye Kokkiz, Research Assistant, Fenerbahce University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020/0072
Record Dates: First submitted 2023-08-16; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Aspiration, Respiratory; Pain; Mucosal Irritation; Infant
MeSH Terms: conditions — Respiratory Aspiration; Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This study was designed as randomized, controlled, and experimental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Positive Pressure Group) (Experimental): The nasopharyngeal suction with positive pressure method was employed in the sample group. In this method, the infant's head is turned to the side, to the nostril on the other side 1-2 ml of physiological saline (PS- Mustela trademark), is injected with a 2,5-milliliter syringe (Can Medikal trademark), and then positive pressure is exerted with the help of the end of the oxygen connection hose (CGR Medikal trademark) from the same nostril, with oxygen or air supply at 5-8 lt/min (liter/minute) (if the baby requires oxygen, using an oxygen source) and the nasopharyngeal secretions are removed from the nostril into which physiological saline (PS) has been not injected. The oxygen connection hose is held one centimeter away from the infant's nostril. The researchers prepared a guideline for nasopharyngeal suction with positive pressure based on the literature.
  Interventions: Device: Experimental group
- Control group (Negative Pressure Group) (Active Comparator): The nasopharyngeal suction with negative pressure method was employed in the control group in this study. In this method, the nasal secretions were softened with 1-2 ml of physiological saline (PS- Mustela trademark) like experimental group, and then negative pressure suction was performed using a pine-tipped suction set (Bıcakcılar trademark). The suction pressure was kept between 60 and 80 mmHg, and no suction lasted for more than 15 seconds
  Interventions: Device: control group

INTERVENTIONS:
Device: Experimental group — THE EFFECTS OF NASOPHARYNGEAL SUCTION POSITIVE PRESSURE
  Arms: Experimental group (Positive Pressure Group)
Device: control group — THE EFFECTS OF NASOPHARYNGEAL SUCTION NEGATIVE PRESSURE
  Arms: Control group (Negative Pressure Group)

SUMMARY:
Objective: The aim of the study is to determine the effects of nasopharyngeal suction with negative and positive pressure on the pain level, respiratory parameters, and mucosal irritation in infants.

Materials and Methods: This study was conducted as a posttest randomised controlled experimental research. The data were collected at XX Training and Research Hospital between January and November 2020. While the positive pressure suction method was applied to the experimental group, the negative pressure suction method was applied to the control group.

DETAILED DESCRIPTION:
Nurses are responsible for suction function to clear the airway from secretions for effective breathing. Suction is defined as the removal of secretions of the respiratory system with a negative pressure vacuum device. In patients who are unable to extract respiratory secretions independently, suction is essential to maintain the oxygen demand and ventilation at the desired level and remove these secretions.

The infant's respiratory and circulatory systems may be adversely affected as a result of the suction procedure, and several complications such as trauma, haemorrhage, and pain may develop. Suction is therefore one of the procedures that should be applied with caution in infants. Suction procedures for the respiratory tract in infants include oro/nasopharyngeal and endotracheal suction and suction methods include open and closed system suction methods.

Oro/nasopharyngeal suction is a method that requires the use of negative pressure to remove secretions from the oropharynx, nasopharynx, or both. When a foreign body penetrates the trachea from the pharynx, when respiratory secretions are too much, or when the secretion cannot be removed by normal cilia movement, coughing holds an important role. Inability to cough leads to atelectasis, pneumonia, and respiratory failure during infection of the respiratory tract. The cough reflex matures around the age of five in children. Adults are able to quickly remove existing airway secretions, but children with excessive airway secretions prior to this age are unable to do so easily. These secretions may be removed through either nasopharyngeal or oropharyngeal suction.

There are several risks and complications associated with suction procedure. The most common are hypoxia, bradycardia, tachycardia, hypotension, hypertension, cardiac arrhythmia, cardiac arrest, atelectasis, bronchospasm, elevated intracranial pressure, nosocomial infection, tracheobronchial damage, and pain. Hypoxemia is the most prevalent and serious complication among them. To avoid the suction-induced hypoxemia, different suction methods are being developed and novel devices are being employed.Suction, a painful procedure, has been reported to negatively impact the physiological parameters, comfort, sleep, growth, and hospital stay of infants. The primary goal of pain management in infants is to minimise the pain experienced by infants due to various medical procedures and allow them to cope with the pain.

When the literature was reviewed, it was observed that the respiratory rate, heart rate, SpO2 and tidal volumes of the patients were assessed as respiratory parameters, while spirometry was utilized to assess respiratory function.

Trauma is another complication of negative pressure suction. Suctioning of the tracheal, oral, and nasopharyngeal mucosa caused by negative pressure may result in haemorrhage and ulceration. As a result of the increased vacuum pressure generated during suction, the mucosal fragments are displaced from the catheter holes and absorbed.

Objective This study aimed to determine the effects of nasopharyngeal suction with negative and positive pressure on the level of pain, respiratory parameters, and mucosal irritation in infants.

Research Hypotheses H0: There is no difference between positive pressure nasopharyngeal aspiration procedure and negative pressure nasopharyngeal aspiration procedure.

H1: The level of pain felt by infants during nasopharyngeal suction with positive pressure is lower than the level of pain they suffer during nasopharyngeal suction with negative pressure.

H2: In infants, the SpO2 level after nasopharyngeal suction with positive pressure is higher than the SpO2 level following nasopharyngeal suction with negative pressure.

H3: In infants, the respiratory rate after nasopharyngeal suction with positive pressure is less affected than the respiratory rate following nasopharyngeal suction with negative pressure.

H4: In infants, the mucosal irritation caused by the nasopharyngeal suction with positive pressure is less than the mucosal irritation caused by the nasopharyngeal suction with negative pressure.

ELIGIBILITY:
Inclusion Criteria:

* Existence of secretion

Exclusion Criteria:

* Being premature
* without family consent

Ages: 37 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-03-11 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Pain | Before the suction procedure 1st minute after the procedure 5st minute after the procedure 15st minute after the procedure
  Determining the pain level with the Wong-Baker Faces Pain Rating Scale. Wong-Baker FACES Pain Rating Scale (Wong & Baker, 1988) is an adaptation of the "Faces Rating Scale" which is a picture projection technique for assessing child pain and utilizes 6 illustrations of faces that a child in pain uses to best describe their present level of pain.
  Face 0 depicts a happy face with no pain. Face 5 depicts a crying face that "hurts as much as you can imagine, although you don't have to be crying to feel this bad." Responses on the 5-point scale range from 0 (very happy, no hurt) to 5 (hurts as much as you can imagine).
Respiratory Parameters | Before the suction procedure 1st minute after the procedure 5st minute after the procedure 15st minute after the procedure
  Determining The Effect of Suction on SpO2 level
Mucosal İrritation | Before the suction procedure 1st minute after the procedure 5st minute after the procedure 15st minute after the procedure
  Determining The Existence of Mucosal İrritation (bleeding or absent)

CONTACTS AND LOCATIONS:
Overall Officials: kokkiz, Study Director — Fenerbahce University
Locations (1):
- Istanbul Medeniyet University Goztepe Hospital, Istanbul, Kadiköy, Turkey (Türkiye)